CLINICAL TRIAL: NCT04524156
Title: COVID-19 : Transcutaneous pO2 and pCO2 as Predictive Factors for Acute Respiratory Destress Syndrome in Patients Affected With SARS-Cov-2
Acronym: COVID-pO2-RAAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P2020/238
Record Dates: First submitted 2020-04-30; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: COVID; Acute Respiratory Distress Syndrome; Endothelial Dysfunction
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Functional Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVIS 19 positive (Active Comparator)
  Interventions: Other: Physiology
- COVID 19 negative (Sham Comparator)
  Interventions: Other: Physiology

INTERVENTIONS:
Other: Physiology — Percutaneous O2 and CO2 partial pressures. A PeriFlux system 5000 (Perimed©, Järfälla, Sweden) will be used to monitor TcpO2 and TcpCO2 tensions by means of a PF 5040 unit and a dual TcpO2/CO2 E5280 electrode. The E5280 electrode, covered by a membrane permeable to oxygen (O2) and carbon dioxide (CO2) heats (44°C) the underlying tissue to maximize gas diffusion through the skin. .
  Pulse Oximeter and hemodynamic parameters Pulse oximeter is a portable device largely used to measure real time finger oxygen saturation (SatO2) and heart rate Blood collection After the above said measurements, a venous blood simple will be realized. Plasma concentration of ACE2, Angiotensin II, Angiotensin 1-7, angiotensin 1-9, CC16, will be measured at the Erasme hospital (ELISA method).

SUMMARY:
The first case of a person infected with SARS-Cov-2 virus can be tracked back on November the 17th, 2019, in China. On March 11, 2020, the World Health Organization (WHO) declared COVID-19 outbreak a pandemic. On April 13, COVID-19 is affecting 210 countries and territories worldwide, about 2 million positive cases have been officially declared along with 115.000 deaths. The real number of infected and deaths is scarily higher, considering that up to 65% people are asymptomatic and thus, not tested.

The percentage of patients with COVID-19 needed for intensive care unit (ICU) varied from 5 to 32% in Wuhan, China. It was up to 9% in Lombardy, Italy. According to available data from Lombardy, 99% of patients admitted to the ICU needed respiratory support (88% invasive ventilation, 11% non invasive ventilation).

The aim of the present investigation is to test the hypothesis whether transcutaneous partial O2 and CO2 pressures may be reliable predictive factors for acute respiratory distress syndrome (ARDS) development in hospitalized clinically stable COVID-19 positive patients and to clarify the role of the Angiotensin Converting Enzyme 2 (ACE2) and its final product, angiotensin 2 (Ang II) in the pathogenesis of this systemic disease.

We also aim to test the hypothesis that plasma concentration of Clara Cell protein (CC16) and surfactant protein D (SPD), which are a biomarkers of acute lung injury, are severely decreased in COVID-19 positive patients and the plasma concentration is related to the severity of lung injury.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV2 infection (PCR positive and/or TDM Imaging)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-04 (Estimated); Primary Completion 2021-09-04 (Estimated); Study Completion 2023-05-04 (Estimated)

PRIMARY OUTCOMES:
Transcutaneous pO2 and pCO2 as predictive factors for respiratory deterioration | 6 months
  To test the prognostic utility of TcpO2 and TcpCO2 for the prediction of COVID19 related lung injury and acute respiratory distress syndrome (ARDS) compared to finger oxygen saturation.
Pneumoproteins CC16 and SDP as predictive factors for respiratory deterioration | 6 months
  To test the prognostic utility of CC16 and SPD in patients with COVID19-related acute lung injury
Diagnostic and prognostic utility of plasma concentration of ACE2, Ang II, Ang 1-7, Ang 1-9 in COVID-19 | 6 months
  To test the hypothesis that plasma concentration of ACE2, AngII, Ang 1-7 and Ang 1-9 are profoundly impaired in COVID-19 and may be predictive factors of clinical deterioration

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Morra, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided